CLINICAL TRIAL: NCT01725295
Title: Neurostructural Integration Technique for Fibromyalgia
Acronym: NST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Professor Geraldine McCarthy, Consultant Rheumatologist, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NST
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia treatment; physical therapy; hydrotherapy
MeSH Terms: conditions — Fibromyalgia | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NST (Experimental): A form of physical therapy to relieve symptoms of fibromyalgia
  Interventions: Other: NST
- Hydrotherapy (Active Comparator): An alternate form of physical therapy to relieve symptoms of fibromyalgia
  Interventions: Other: Hydrotherapy

INTERVENTIONS:
Other: NST — A form of physical therapy
  Arms: NST
Other: Hydrotherapy
  Other Names: A form of physical therapy
  Arms: Hydrotherapy

SUMMARY:
Fibromyalgia is a common cause of widespread musculoskeletal pain. The investigators have found that our patients seem to benefit from a soft tissue physical therapy called neurostructural integration therapy (NST). The purpose of this study was to compare NST to hydrotherapy which is already used to manage fibromyalgia symptoms.

DETAILED DESCRIPTION:
Twenty female patients who met the American College of Rheumatology diagnostic criteria for the classification of FM were enrolled in the study. Patients were randomly allocated to receive either hydrotherapy or NST. Patient evaluations were performed at baseline, six weeks, three months, and six months. Primary outcome measures included the SF-36 quality of life questionnaire, the Fibromyalgia Impact Questionnaire and the Total Myalgic Score. Duration of morning stiffness and duration of weekly aerobic exercise as reported by the participants were secondary outcome measures. Statistics analysis was performed by standard parametric and non parametric methods.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who fulfills ACR diagnostic criteria for fibromyalgia

Exclusion Criteria:

* Patients with established ischemic heart disease, uncontrolled hypertension or diabetes, hypothyroidism, severe depression

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Misericordiae Hospital, Dublin, Dublin, Ireland